CLINICAL TRIAL: NCT04820699
Title: Comparative Study of Post Isometric Relaxation and Mulligan Bent Leg Raise on Hamstring Tightness in High School Students
Brief Title: Post Isometric Relaxation and Mulligan Bent Leg Raise on Hamstring Tightness in High School Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/18/1008
Record Dates: First submitted 2021-03-26; First posted 2021-03-29 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Hamstring Injury; Hamstring Tendon Injury

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- post isometric relaxation (Experimental): Group A received Post isometric relaxation technique (MET).The participants performed isometric contractions using 20% of their strength, 5 second holds with 5 seconds rest time in between each contraction
  Interventions: Other: post isometric relaxation and muligan bent leg raise
- mulligan bent leg raise (Experimental): Group B: Mulligan bent leg raise technique. Isometric contraction of hamstring muscle for progressively five greater position of hip flexion; three pain-free repetitions with 5 second hold was performed by participants
  Interventions: Other: muligan bent leg raise

INTERVENTIONS:
Other: post isometric relaxation and muligan bent leg raise — 6 week intervention
  Arms: post isometric relaxation
Other: muligan bent leg raise — muligan bent leg raise
  Arms: mulligan bent leg raise

SUMMARY:
This project was a Randomized clinical trial conducted COMPARATIVE STUDY OF POST ISOMETRIC RELAXATION AND MULLIGAN BENT LEG RAISE ON HAMSTRING TIGHTNESS IN HIGH SCHOOL STUDENTS

DETAILED DESCRIPTION:
Non Probability Convenient sampling was done. Patients following eligibility criteria from high schools located in vicinity of Jhang district were considered. Sample size was calculated with Epitool calculator. 28 Participants were randomly allocated in two groups equally via convenient sampling method. Baseline assessment was done initially. Group A was given post isometric relaxation and Group B was given mulligan bent leg raise Duration of research was almost 6 months. All 28 involved subjects were given 12 treatment sessions over a six-week period, which consisted of 02 treatment sessions per week . Then tightness of hamstrings was assessed by AKET, SLR and FTF test. The baseline outcome measures consisted of pain assessment using Numeric rating scale (NPRS), knee joint goniometry in active knee extension test (AKET) and straight leg raise (SLR), modified finger to floor test (FTF) to assess the flexibility of hamstring muscles. . All participants were provided written informed consent prior to commencement of the procedures. Data was analyzed by using SPSS version 23.

ELIGIBILITY:
Inclusion Criteria:

Asymptomatic Individuals of both gender, aged 13 to 18 years were evaluated for unilateral or bilateral Hamstring tightness. Those who were unable to reach more than 160 degree of knee extension with hip held at 90 degree of flexion, as measured with the thigh held at 90 degrees of hip flexion), unable to complete SLR and meet the criteria of finger to floor test

were included.

Exclusion Criteria:

Individuals were excluded who presented with previous injury of lower limb or pain duration of one year. Also any deformities related to spine, hip and knees or any neurological disorder or with history of lower limb fracture or surgery were also excluded.Subjects with hamstring tightness associated with muscle soreness or with Inflammatory condition that could affect motion were also exluded from the study

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-08-15 (Actual)

PRIMARY OUTCOMES:
NUMERIC PAIN RATING SCALE for pain | 2 months
  0-10 Rating,0 means no pain and 10 severe pain
Knee joint goniometry in active knee extension test (AKET) | 2 months
  The 90/90 test, also known as the Active Knee Extension (AKE) Hamstring Flexibility Test, measures hamstring flexibility, particularly when the hip is flexed. purpose: to assess the range of active knee extension in a position of hip flexion, as required in running and kicking.
straight leg raise (SLR) test | 2 months
  If symptoms are primarily back pain, it is most likely the result of a disc herniation applying pressure on the anterior theca of the spinal cord, or the pathology causing the pressure is more central. "Back pain only" patients who have a disc prolapse have smaller, more central prolapses.[1] If pain is primarily in the leg, it is more likely that the pathology causing the pressure on neurological tissue(s) is more lateral.[1] Disc herniations or pathology causing pressure between the two extremes are more likely to cause pain in both areas.
modified finger to floor test (FTF) | 2 months
  If the FTF test is limited by pain, the location and pain score out of 10 should be should be documented. If the FTF test is 0cm or the patient is able to place their palms to the floor with no pain, 10 with maximum pain

CONTACTS AND LOCATIONS:
Overall Officials: warda saleem, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah IU, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalanekar TA, Koley S. A Comparative Study of Mulligans Bent Leg Raise versus Muscle Energy Technique in Asymptomatic Individuals with Hamstring Tightness.